CLINICAL TRIAL: NCT03417011
Title: FORWARD PRO Study Interventional Post-market Study With the Evolut™ PRO System
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT17050EVR003
Record Dates: First submitted 2018-01-18; First posted 2018-01-31 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Medtronic CoreValve™ Evolut™ PRO System (Evolut™ PRO System) — Transcatheter Aortic Valve Replacement with Medtronic Evolut PRO system

SUMMARY:
Prospective, single-arm, multi-center, interventional post-market study. After signing informed consent, eligible subjects will be implanted with the CE marked Evolut™ PRO system.

The investigation purpose is to evaluate the acute and long term clinical performance and safety of Evolut™ PRO in a routine hospital setting in patients with symptomatic native aortic valve stenosis or a stenosed, insufficient, or combined surgical bioprosthetic valve failure necessitating valve replacement within the approved intended use in local geography.

DETAILED DESCRIPTION:
Approximately 600 subjects implanted with the Evolut™ PRO at up to 40 sites in Europe. Other regions may be added depending on the regulatory status of the device.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic native aortic valve stenosis or a stenosed, insufficient, or combined surgical bioprosthetic valve failure necessitating valve replacement
* High or greater risk for surgical aortic valve replacement as estimated by the heart team OR, 75 years or older and at intermediate risk for surgical AVR (STS risk score ≥4% or with an estimated hospital mortality ≥4% as assessed by the heart team)
* Acceptable candidate for treatment with the Evolut™ PRO system in conformity with the Instructions for Use and the local regulations
* Able and willing to return to the implanting site at the following follow-up visits: 1-year, 3-year and 5-year
* Written informed consent obtained without assistance from a legal representative prior to enrollment in the study.

Exclusion Criteria:

* Known hypersensitivity or contraindication to aspirin, heparin (HIT/HITTS) and bivalirudin, ticlopidine, clopidogrel, Nitinol (Titanium or Nickel), or sensitivity to contrast media, which cannot be adequately premedicated
* Preexisting mechanical heart valve in aortic position
* Ongoing sepsis, including active endocarditis
* Anatomically not suitable for the Evolut™ PRO system
* Estimated life expectancy of less than 1 year
* Participating in another trial that may influence the outcome of this study
* Need for emergency surgery for any reason
* Inability to understand and respond to the quality of life questionnaire

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with symptomatic native aortic valve stenosis or a stenosed, insufficient, or combined surgical bioprosthetic valve failure necessitating valve replacement within the approved intended use in local geography.
Sampling Method: Non-Probability Sample
Enrollment: 638 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2024-02-26 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | 30 days post procedure
  The all-cause mortality rate at 30 days post procedure meets a prespecified performance goal of 5.5%.

SECONDARY OUTCOMES:
Total AR | 24 hours to 7 days post procedure (prior to discharge)
  The percentage of subjects graded as none or trace total aortic regurgitation at discharge is greater than a prespecified performance goal of 67.1%.
VARC-2 composite safety endpoint | through 5 years from enrollment until end of study
  Event rate of the VARC-2 composite safety endpoint through 5 years from enrollment until end of study, which includes the following components:
  * All-cause mortality
  * All stroke (disabling and non-disabling)
  * Life-threatening bleeding
  * Acute kidney injury: stage 2 or 3 (including renal replacement therapy)
  * Coronary artery obstruction requiring intervention
  * Major vascular complication
  * Valve-related dysfunction requiring repeat procedure (BAV, TAVI, or SAVR)
Individual components of the VARC-2 composite safety endpoint | through 5 years from enrollment until end of study
  Event rates of the individual components of the VARC-2 composite safety endpoint through 5 years until end of study
Rate of new permanent pacemaker implant | 30 days post procedure
  Rate of new permanent pacemaker implant at 30 days post procedure
Device success rate | 24 hours to 7 days post procedure (prior to discharge)
  Device success rate at 24 hours to 7 days post procedure (prior to discharge), defined according to the VARC-2 guidelines as:
  * Absence of procedural mortality, AND
  * Correct positioning of a single prosthetic heart valve into the proper anatomical location, AND
  * Intended performance of the prosthetic heart valve, defined as the absence of patient prosthesis mismatch and mean gradient <20 mmHg (or peak velocity <3 m/sec), AND
  * No moderate or severe prosthetic valve regurgitation.
Hemodynamic performance | 24 hours to 7 days (prior to discharge), 1-year, 3-year and 5-year post
  Hemodynamic performance at 24 hours to 7 days (prior to discharge), 1-year, 3-year and 5-year post procedure, including the mean prosthetic valve gradient as measured by transthoracic echocardiography (TTE) and assessed by an independent core laboratory.
Hemodynamic performance | 24 hours to 7 days (prior to discharge), 1-year, 3-year and 5-year post
  Hemodynamic performance at 24 hours to 7 days (prior to discharge), 1-year, 3-year and 5-year post procedure, including the effective orifice area as measured by transthoracic echocardiography (TTE) and assessed by an independent core laboratory.
Hemodynamic performance | 24 hours to 7 days (prior to discharge), 1-year, 3-year and 5-year post
  Hemodynamic performance at 24 hours to 7 days (prior to discharge), 1-year, 3-year and 5-year post procedure, including the degree of prosthetic valve regurgitation (transvalvular, paravalvular and total) as measured by transthoracic echocardiography (TTE) and assessed by an independent core laboratory.
Change in NYHA functional status | From baseline to 30-day, 1-year, 3-year, and 5-year post procedure
  Change in NYHA functional status from baseline to 30-day, 1-year, 3-year, and 5-year post procedure
Change in Quality of Life score | From baseline to 30-day, and 1-year, 3-year, and 5-year post procedure
  Change in Quality of Life score (EQ-5D questionnaire) from baseline to 30-day, and 1-year, 3-year, and 5-year post procedure. The EQ-5D descriptive system comprises five dimensions and each dimension has five levels of severity. The subject is asked to indicate his/her health state by ticking (or placing a cross) in the box against the most appropriate statement in each of the five dimensions. The EQ VAS records the subject's self-rated health on a 20 cm vertical, visual analogue scale. The subject marks an X on the scale to indicate how his/her health is TODAY and then writes the number they marked on the scale in the box below.

CONTACTS AND LOCATIONS:
Locations (39):
- LKH - Universitätsklinikum, Graz, Austria
- Belgium (2):
  - Universitair Ziekenhuis Antwerpen, Antwerp
  - CHU de Liège - Hôpital du Sart Tilman, Liège
- Rigshospitalet, Copenhagen, Denmark
- Turun Yliopistollinen Keskussairaala, Turku, Finland
- France (3):
  - CHU Bordeaux, Bordeaux
  - Hôpital Henri Mondor, Créteil
  - Clinique Pasteur, Toulouse
- Germany (11):
  - Herz- und Diabeteszentrum NRW - Ruhr-Universität Bochum, Bad Oeynhausen
  - Deutsches Herzzentrum Berlin, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Sana-Herzzentrum Cottbus GmbH, Cottbus
  - Herzzentrum Dresden GmbH Universitätsklinik, Dresden
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Essen, Essen
  - Asklepios Klinik St. Georg, Hamburg
  - Herzzentrum Leipzig GmbH, Leipzig
  - Deutsches Herzzentrum München Klinik an der TU München, Munich
  - SANA Herzchirurgie Stuttgart GmbH, Stuttgart
- Israel (2):
  - Hadassah Medical Organisation, Jerusalem
  - Rabin Medical Center - Beilinson Hospital, Petah Tikva
- Italy (5):
  - Azienda Ospedaliera Spedali Civili di Brescia, Brescia
  - AOU Presidio Gaspare Rodolico Policlinico, Catania
  - Azienda Ospedaliera Ospedale Niguarda Cà Granda, Milan
  - IRCCS Policlinico San Donato, Milan
  - Azienda Ospedaliero Universitaria Pisana - Stabilimento di Cisanello, Pisa
- Netherlands (3):
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Catharina Ziekenhuis Eindhoven, Eindhoven
  - Erasmus Medisch Centrum, Rotterdam
- Oslo Universitetssykehus-Ullevål, Oslo, Norway
- University Medical Centre, Ljubljana, Slovenia
- Spain (3):
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Central de Asturias, Oviedo
  - Complejo Hospitalario Universitario de Santiago de Compostela, Santiago de Compostela
- Switzerland (2):
  - Inselspital - Universitätsspital, Bern
  - Universtitätsspital Zürich, Zurich
- United Kingdom (3):
  - Royal Victoria Hospital - Belfast Health and Social Care Trust, Belfast
  - St. George's Hospital, London
  - The Royal Wolverhampton Hospitals NHS - New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Van Mieghem NM, Windecker S, Manoharan G, Lancellotti P, Tamburino C, Kornowski R, Thiele H, Danenberg H, Fiorina C, Scholtz W, Brecker S, Ruge H, Opdahl A, Amoroso G, Bedogni F, Petronio AS, Nickenig G, Harnath A, Kempfert J, Oh JK, Eisenberg RE, Grube E. Three-Year Outcomes With a Supra-Annular, Self-Expanding Bioprosthesis and a Pericardial Wrap-The FORWARD PRO Study. Catheter Cardiovasc Interv. 2025 Feb;105(3):577-587. doi: 10.1002/ccd.31335. Epub 2024 Dec 16. PMID 39686582
- [Derived] Manoharan G, Grube E, Van Mieghem NM, Brecker S, Fiorina C, Kornowski R, Danenberg H, Ruge H, Thiele H, Lancellotti P, Sondergaard L, Tamburino C, Oh JK, Fan Y, Windecker S. Thirty-day clinical outcomes of the Evolut PRO self-expanding transcatheter aortic valve: the international FORWARD PRO study. EuroIntervention. 2020 Nov 20;16(10):850-857. doi: 10.4244/EIJ-D-20-00279. PMID 32748789